CLINICAL TRIAL: NCT02335658
Title: Long-term Study of DSP-5423P in Patients With Schizophrenia <Phase 3>
Brief Title: Long-term Study of DSP-5423P in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4904040; JapicCTI-152765 (Registry Identifier: JAPIC Clinical Trials Informaton)
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSP-5423P (Experimental): Percutaneous
  Interventions: Drug: DSP-5423P

INTERVENTIONS:
Drug: DSP-5423P — 40-80mg/day

SUMMARY:
The study evaluates the long term safety of DSP-5423P in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have schizophrenia diagnosed by DSM-5, diagnostic criteria
* Patients who are aged 18 years or older at informed consent
* Patient understands the objectives and procedures of the study and who provide written voluntarily consent to participate in the study, etc.

Exclusion Criteria:

* Patients who fall under a contraindication listed in the LONASEN® package insert
* Patients with Parkinson disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (1):
- 38 Sites, Tokyo, Japan

REFERENCES:
- [Derived] Iwata N, Ishigooka J, Naoi I, Matsumoto M, Kanamori Y, Nakamura H, Higuchi T. Long-Term Safety and Efficacy of Blonanserin Transdermal Patches in Japanese Patients with Schizophrenia: A 52-Week Open-Label, Multicenter Study. CNS Drugs. 2020 Jan;34(1):103-116. doi: 10.1007/s40263-019-00692-6. PMID 31883082

RESULTS

PARTICIPANT FLOW:
Groups:
- DSP-5423P (Cohort 1): Percutaneous DSP-5423P: 40-80mg/day, once daily The initial dose of DSP-5423P in Cohort 1 was corresponding to the final dose of DSP-5423 (tablet) in previous period.
- DSP-5423P (Cohort 2): Percutaneous DSP-5423P: 40-80mg/day, once daily The initial dose of DSP-5423P in Cohort 2 was 40 mg/day
Period: Overall Study
Arm/Group | DSP-5423P (Cohort 1) | DSP-5423P (Cohort 2)
Started | 97 (97 subjects in Cohort 1 and 103 subjects in Cohort 2 started to receive DSP-5423P.) | 103
Completed | 57 (57 subjects in Cohort 1 and 59 subjects in Cohort 2 completed the study.) | 59
Not Completed | 40 | 44
Not completed — Adverse Event | 18 | 12
Not completed — Lack of Efficacy | 4 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 13 | 21
Not completed — non-compliance | 2 | 3
Not completed — other reason | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety population-received at least one dose of study medication
Groups:
- DSP-5423P (Cohort 1); DSP-5423P (Cohort 2): Percutaneous
  DSP-5423P: 40-80mg/day
- Total: Total of all reporting groups
Arm/Group | DSP-5423P (Cohort 1) | DSP-5423P (Cohort 2) | Total
Number analyzed (Participants) | 97 | 103 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (14.43) | 43.6 (12.63) | 43.8 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 97 | 103 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 97 | 103 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 97 | 103 | 200

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events and Adverse Drug Reactions, Etc.
Description: Number of Subjects With Adverse Event (AE) and Adverse Drug Reaction (ADR) An adverse event (AE) is any untoward medical occurrence in a study subject administered a medicinal (investigational) product and which does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease occurring after the administration of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
  An adverse drug reaction (ADR) is any AE which has a causal relationship with this treatment.
Time Frame: week 52
Population: Safety population-received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Groups:
- DSP-5423P (Overall): Percutaneous
  DSP-5423P: 40-80mg/day
Arm/Group | DSP-5423P (Cohort 1) | DSP-5423P (Cohort 2) | DSP-5423P (Overall)
Number analyzed (Participants) | 97 | 103 | 200
Participants
  Subjects with any AE | 82 | 92 | 174
  Subjects with any treatment-related ADR | 60 | 77 | 137

2. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week52 and Week 52 Last Observation Carried Forward(LOCF) From DSP-5423P Baseline
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and 3 subscales: the Positive subscale assesses hallucinations, delusions, and related symptoms; the Negative subscale assesses emotional withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
  The LOCF endpoint is defined as the last data captured on Day 1 through 7 days after the final application of DSP-5423P.
Time Frame: Week 52, Week 52 (LOCF)
Population: Safety population-received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSP-5423P (Cohort 1) | DSP-5423P (Cohort 2)
Number analyzed (Participants) | 97 | 103
units on a scale
  Baseline | 63.6 (21.23) | 67.5 (21.34)
  Change at Week 52 | -3.5 (8.41) | -9.2 (15.08)
  Change at Week 52 (LOCF) | -0.1 (11.59) | -3.4 (15.30)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 52 weeks.
Groups:
- DSP-5423P (Overall): Percutaneous
  DSP-5423P: 40-80mg/day
  Cohort 1 + Cohort 2
Arm/Group | DSP-5423P (Cohort 1) | DSP-5423P (Cohort 2) | DSP-5423P (Overall)
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/103 | 0/200
Serious Adverse Events (participants affected / at risk) | 6/97 | 6/103 | 12/200
Other Adverse Events (participants affected / at risk) | 82/97 | 92/103 | 174/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSP-5423P (Cohort 1) (N=97) | DSP-5423P (Cohort 2) (N=103) | DSP-5423P (Overall) (N=200)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 2 (2) | 4 (4) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSP-5423P (Cohort 1) (N=97) | DSP-5423P (Cohort 2) (N=103) | DSP-5423P (Overall) (N=200)
Hyperprolactinaemia (Endocrine disorders) | 7 (8) | 7 (7) | 14 (15)
Dental caries (Gastrointestinal disorders) | 5 (7) | 8 (9) | 13 (16)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (7) | 10 (12)
Vomiting (Gastrointestinal disorders) | 7 (8) | 3 (4) | 10 (12)
Application site dermatitis (General disorders) | 8 (8) | 2 (9) | 10 (17)
Application site erythema (General disorders) | 18 (23) | 27 (38) | 45 (61)
Application site pruritus (General disorders) | 9 (9) | 14 (14) | 23 (23)
Nasopharyngitis (Infections and infestations) | 29 (42) | 33 (46) | 62 (88)
Blood prolactin increased (Investigations) | 2 (2) | 12 (13) | 14 (15)
Weight increased (Investigations) | 3 (3) | 7 (7) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 13 (13)
Akathisia (Nervous system disorders) | 6 (6) | 14 (18) | 20 (24)
Headache (Nervous system disorders) | 6 (7) | 1 (1) | 7 (8)
Tremor (Nervous system disorders) | 4 (4) | 10 (11) | 14 (15)
Insomnia (Psychiatric disorders) | 7 (7) | 11 (11) | 18 (18)
Schizophrenia (Psychiatric disorders) | 7 (7) | 5 (7) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02335658/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT02335658/SAP_001.pdf